CLINICAL TRIAL: NCT01762254
Title: Prospective Randomized Trial of Incisionless Versus Conventional Laparoscopic Colectomy for Left-sided Colonic Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Cheung Yui Shan, Department of Surgery, Pamela Youde Nethersole Eastern Hospital, Pamela Youde Nethersole Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKEC-2009-023
Record Dates: First submitted 2012-11-29; First posted 2013-01-07 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Pain,; Postoperative Wound Complication
Keywords: pain score; complication
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- incisionless laparoscopic colectomy (Active Comparator): incisionless laparoscopic colectomy: Laparoscopic colectomy is being performed in the same manner as conventional laparoscopic colectomy, except that at the end of procedure, the TEO device with the outer diameter of 4cm is inserted into the anus for the delivery of specimen and insertion of anvil instead of creating a small wound as in the conventional laparoscopic colectomy. Finally, intra-corporeal anastomosis is performed in the same manner with the TEO device removed.
  Interventions: Procedure: incisionless laparoscopic colectomy
- conventional laparoscopic colectomy (Active Comparator): conventional laparoscopic colectomy: The operation is completed by laparoscopic instruments using video laparoscopy. At the end of the procedure, pneumoperitoneum is abolished and a small wound was created for the delivery of bowel and insertion of anvil of the circular stapler. Finally, pneumoperitoneum is re-created for intra-corporeal anastomosis
  Interventions: Procedure: conventional laparoscopic colectomy

INTERVENTIONS:
Procedure: incisionless laparoscopic colectomy — Arm 1:Incisionless Laparoscopic Colectomy Laparoscopic colectomy is being performed in the same manner as conventional laparoscopic colectomy, except that at the end of procedure, the TEO device with the outer diameter of 4cm is inserted into the anus for the delivery of specimen and insertion of anvil instead of creating a small wound as in the conventional laparoscopic colectomy. Finally, intra-corporeal anastomosis is performed in the same manner with the TEO device removed.
  Arms: incisionless laparoscopic colectomy
Procedure: conventional laparoscopic colectomy — Arm 2: Conventional Laparoscopic colectomy The operation is completed by laparoscopic instruments using video laparoscopy. At the end of the procedure, pneumoperitoneum is abolished and a small wound was created for the delivery of bowel and insertion of anvil of the circular stapler. Finally, pneumoperitoneum is re-created for intra-corporeal anastomosis
  Arms: conventional laparoscopic colectomy

SUMMARY:
To compare the two surgical options in their short-term and long term outcomes in the management of early left-sided colorectal cancers. The hypothesis is that the incisionless approach will result in less postoperative pain and wound related complications.

DETAILED DESCRIPTION:
For the left-sided colorectal cancer, the investigators performed colectomy with primary anatomosis. Currently the investigators have two methods of minimal access approach to the abdominal cavity in order to complete this operation:

1. Conventional Laparoscopic colectomy The operation is completed by laparoscopic instruments using video laparoscopy. At the end of the procedure, pneumoperitoneum is abolished and a small wound was created for the delivery of bowel and insertion of anvil of the circular stapler. Finally, pneumoperitoneum is re-created for intra-corporeal anastomosis
2. Incisionless Laparoscopic Colectomy Laparoscopic colectomy is being performed in the same manner as conventional laparoscopic colectomy, except that at the end of procedure, the Transanal Endoscopic Operation (TEO) device with the outer diameter of 4cm is inserted into the anus for the delivery of specimen and insertion of anvil instead of creating a small wound as in the conventional laparoscopic colectomy. Finally, intra-corporeal anastomosis is performed in the same manner with the TEO device removed.

These two operations are essentially identical except for the surgical access for the delivery of specimen and insertion of anvil. Laparoscopic colectomy and the use of Transanal Endoscopic Operation(TEO)device have been practiced in the United States and Europe for over 10 years. Large scale studies in the literature have demonstrated the safety and benefits of laparoscopic colectomy for colonic tumors and the oncological outcomes have not shown to be inferior to open approach. With the use of TEO device, the investigators can perform laparoscopic colectomy without abdominal incision for those early left-sided colonic tumors and thus it can eliminate the wound-related complications theoretically. In order to find out which one is a better procedure, the investigators are carrying out a clinical trial to compare the two surgical options in their short-term and long term outcomes.The results of this study may have an impact on the care of similar patients in the future.

ELIGIBILITY:
Inclusion Criteria:

patients >18 years old and diagnosed to have operable left-sided colorectal cancers distal to the splenic flexure and proximal to the upper rectum were potential candidates.

Exclusion Criteria:

1. Patient who did not give informed consent;
2. Patient who were considered unfit for operative treatment;
3. Patient presented as acute surgical emergencies, including intestinal obstruction, peritonitis, or pericolic abscess, etc.;
4. Patients with metastatic diseases on preoperative work up;
5. Patient with synchronous tumours or polyps which necessitate extended or additional resection;
6. Patients with large bulky tumor as demonstrated on preoperative colonoscopy or computed tomography showing serosal involvement or invasion to contiguous organs.
7. Patients with anal stenosis that precluded the insertion of TEO device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pain score | average of 1 week
  participants will be followed for the pain score during the duration of hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
wound complication | up to 30 days after the operation
  The patient will be followed for up to 30 days after the operation or till occurrence of event

OTHER OUTCOMES:
intraoperative blood loss | From the start of operation till operation finished
  From the start of operation till operation finished
operative time | From the start of operation till operation finished
  From the start of operation till operation finished
length of hospital stay | From the date after operation to date of discharge,an expected average of within 1 week
  From the date after operation to date of discharge,an expected average of within 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Yui Shan Cheung, FRACS, Principal Investigator — Department of Surgery, Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Department of Surgery, Pamela Youde Nethersole Eastern Hospital, Hong Kong, China